CLINICAL TRIAL: NCT06874764
Title: Effects of Agility and Cognitive Training With Reaction System on Cognitive Functions and Walking in Individuals With Multiple Sclerosis
Brief Title: Effect of Training With Wireless Lightning Reaction Systems on Cognitive Functions in Individuals With Multiple Sclerosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yunus Emre Meydanal, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 25-5/4
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Cognitive; Virtual reality; Agility; Training; Gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The intervention group will be trained with a difficulty appropriate to their individual levels for 2 months using the reaction system 2 days a week to improve agility and cognitive functions, and if the participant can easily perform the relevant training, the difficulty will be increased by one level. Agility training aims to reach the light side sensor with the hand in order and to do this within the specified time, and aims to speed up the participant's reaction time in the foreground. Cognitive training consists of different trainings such as finding the different image illuminated in 8 sensors, finding two identical signs, remembering the order in which the sensors light up, and touching the sensors in that order. These trainings aim to increase the participant's quick thinking and decision making, and to improve attention, visual memory, visual processing speed, and cognitive functions. Each training session will last approximately 30 minutes.
  Interventions: Other: Wireless Lighting Reaction System Training(Agility plus Cognitive)
- Control Group (No Intervention): The control group will not receive any intervention. They will be asked to continue their normal lives.

INTERVENTIONS:
Other: Wireless Lighting Reaction System Training(Agility plus Cognitive) — Agility training and Cognitive trainings(cognitive trainings ready within the device: Eye for detail, Hawk eye, Juggle Factor)
  Arms: Training Group

SUMMARY:
When the literature is examined, balance disorders, walking disorders and cognitive problems are frequently observed in Multiple Sclerosis(MS) patients. Using technologically supported equipment such as reaction systems, cognitive function measurements have been successfully performed in the elderly, and improvements in reaction times have been detected in athletes when used for training purposes. The primary aim of the study is to provide improvement in agility and cognitive functions in patients using a technology-supported reaction device. In addition, it aims to improve balance function assessed with static posturography and gait parameters assessed with gait analysis by increasing sensory input and shortening reaction time. As a result of the agility and cognitive training performed, we aim to provide improvement in MS-related quality of life and decrease in disability.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an immune-mediated central nervous system disease characterized by inflammation, demyelination, and axonal damage. Myelin sheaths, oligodendrocytes, and to a lesser extent the axon and the nerve cell itself are damaged.Balance problems can be seen even in the early stages of MS. In the later stages of the disease, they are the primary cause of falls. Balance is defined as the body's ability to maintain its center of gravity with minimal sway. Approximately two-thirds of MS patients report balance or coordination problems that affect their daily lives.Gait impairment is common in MS patients. Walking speed, quality and endurance are the components of the Expanded Disability Status Scale (EDSS), which is most commonly used to monitor MS-related disability and disease progression.Inflammation and demyelination that develop during the MS process have significant effects on central nervous system functions, especially cognitive performance. Approximately 40-70% of people with multiple sclerosis have cognitive impairments such as slowed processing speed, impaired learning and memory functions, and deficits in executive functions. These symptoms affect patients' emotional well-being, work capacity, and quality of life (QoL).Reaction systems (Witty SEM, Microgate, Bolzano, Italia) are devices with computer-aided wireless lighting feature that evaluate and train various visual, cognitive and sensory-motor skills. It consists of an light emitting diode(LED) screen that displays different colors, numbers and characters. This technology is used for evaluation and special training for reactivity, agility and coordination.A total of 40 male and female individuals between the ages of 18-55 will be included in the study. Participants will be divided into two different groups as intervention and control in equal numbers. In both groups, the Brief International Cognitive Assessment for MS (BICAMS) battery, Berg Balance Scale, Hospital Anxiety and Depression Scale (HADS), Fatigue Severity Scale (FSS) and Short Form-36 (SF-36) health questionnaire will be applied to the participants before the study. BICAMS is a battery consisting of the California Verbal Learning Test II (CVLT II), Symbol Digit Modalities Test (SDMT) and Brief Visuospatial Memory Test-Revised (BVMTR) subscales used in the assessment of cognitive status in MS patients.In both groups, before the study, static posturography (HUR SMART BALANCE BTG4) will be used and the patients' balance-related measurements such as forward-backward and sideways swings, swing speeds during pressure, and measurements of the static balance scores provided by the device will be noted, respectively, in the eyes open normal ground - eyes closed normal ground - eyes open soft mat - eyes closed soft mat ground.In addition, using the pressure-gait analysis system (DIERS International GmbH, Schlangenbad, Germany), the participants will undergo pressure analysis and walking evaluation on a treadmill at a walking speed chosen by the patient between 2-5 km/h for approximately 20 seconds.The intervention group will be trained at a difficulty level appropriate to their individual levels to improve agility and cognitive functions using the reaction system 2 days a week for 2 months, and if the participant can easily perform the relevant training, the difficulty will be increased by one level. Each training session will last approximately 30 minutes. There will be no intervention in the control group. At the end of the 8 weeks, the scales, questionnaires and measurements made before the study will be repeated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-55
* Having a definite MS diagnosis according to the 2017 McDonald criteria.
* EDSS score of 4 or below
* Being able to communicate (speaking and understanding Turkish, no speech disorders)

Exclusion Criteria:

* Regular exercise in the last 6 months
* Having an MS attack in the last month
* Having an MS attack during the study period
* Presence of additional accompanying neurological diseases
* Use of dalfampridine
* Use of antipsychotic and psychostimulant drugs
* Drug and alcohol addiction
* Pregnancy, breastfeeding
* No chronic systemic disease preventing exercise
* Patients who cannot reach the targeted exercise level

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive Functions | 8th week
  the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) is a battery with demonstrated validity and reliability in Turkish, consisting of the California Verbal Learning Test II (CVLT II), Symbol Digit Modalities Test (SDMT) and Brief Visuospatial Memory Test-Revised (BVMTR) subscales, used to assess cognitive status in MS patients SDMT: There is no lower or upper limit for scoring. A higher number of correct answers (higher scores) is associated with better results.
  CVLTII:The upper limit for scoring is 80. A higher number of correct answers (higher scores) is associated with better results.
  BVMTR:The score range is 0-12. Higher scores are associated with better outcomes.

SECONDARY OUTCOMES:
Balance assessment | 8th week
  Berg Balance Scale: It is a scale consisting of 14 tests that measure the ability to maintain balance during different positions, postural changes and movement. The evaluation is based on the person's ability to perform each test independently and/or for a certain time or distance. The rating is made between 0 and 4 points (0: cannot do, 4: normal performance). The total score varies between 0 (dependent) and 56 (independent). High scores are associated with independent movement and low risk of falling. The validity and reliability of this scale has been shown in Turkish.
Anxiety and Depression Status | 8th week
  HADS (Hospital Anxiety and Depression Scale): The scale is a self-report scale. It consists of 14 items, 7 of which investigate depression and 7 of which investigate anxiety symptoms. Responses are evaluated in a four-point Likert format and are scored between 0-3. It is often used for screening purposes. The scale can also be used to evaluate the change in the patient's emotional state. The score range for both subscales are 0-21 High scores indicate an increase in depression and/or anxiety.
Fatigue Assessment | 8th week
  FSS (Fatigue Severity Scale): A nine-item scale designed to assess fatigue as a symptom of various chronic conditions and disorders. The scale addresses the effects of fatigue on daily functioning, questions its relationship to motivation, physical activity, work, family and social life, and asks participants to rate how easily they tire and the extent to which this causes problems for them. Participants respond to nine statements about fatigue on a scale ranging from 1 ("completely disagree") to 7 ("completely agree"). The score range for the test is 9-63. Higher scores on the scale indicate more severe fatigue.FSS measures the severity of fatigue and is widely used in multiple sclerosis patients. The validity and reliability of this scale in Turkish has been demonstrated.
MS Quality of Life | 8th week
  SF-36 (Short Form 36): The SF-36 is a set of general, consistent, and easily administered quality of life measures. These measures are based on patient self-report. The SF-36 has eight subscales; scores are weighted sums of questions in each section, ranging from 0 to 100. Higher scores are associated with better quality of life. Validity and reliability have been demonstrated in Turkish
Static Posture Assessment(Static Balance) | 8th week
  Static Posturography: Static posturography is based on the principle of measuring changes in the center of pressure on a stationary platform. In a calm posture, the body is normally held upright and the center of mass is elevated above the base of support provided by the feet. Although it is generally assumed that the center of pressure (COP) indicates the location of the body's center of mass, discrepancies between the two occur, especially during rapid or high-frequency components of movement.
  Static Balance Score: indicates the individual's ability to stand still with eyes open on a firm surface. It will be calculated automatically by the device and used as a reference for other measurements. Scoring ranges from 0 to 100. Higher scores are associated with better outcomes.
Static Posture Assessment(Visual Dependency) | 8th week
  Static Posturography: Static posturography is based on the principle of measuring changes in the center of pressure on a stationary platform. In a calm posture, the body is normally held upright and the center of mass is elevated above the base of support provided by the feet. Although it is generally assumed that the center of pressure (COP) indicates the location of the body's center of mass, discrepancies between the two occur, especially during rapid or high-frequency components of movement.
  Visual Dependency Score: Visual Dependency Score indicates how closing the eyes can affect an individual's ability to stand still on a firm surface.With eyes closed, the effects of vision on balance are assessed.The score will be calculated automatically by the device. Scoring ranges from 0 to 100. Higher scores are associated with better outcomes.
Static Posture Assessment(Proprioception Disturbance) | 8th week
  Static Posturography: Static posturography is based on the principle of measuring changes in the center of pressure on a stationary platform. In a calm posture, the body is normally held upright and the center of mass is elevated above the base of support provided by the feet. Although it is generally assumed that the center of pressure (COP) indicates the location of the body's center of mass, discrepancies between the two occur, especially during rapid or high-frequency components of movement.
  Proprioception Disturbance Score:indicates how much standing on a soft foam surface can affect the individual's ability to stand still with eyes open.With eyes open and on soft ground, rubber pads restrict the somatosensory system.The score will be calculated automatically by the device. Scoring ranges from 0 to 100. Higher scores are associated with better outcomes.
Static Posture Assessment(Vestibular Dominant) | 8th week
  Static Posturography: Static posturography is based on the principle of measuring changes in the center of pressure on a stationary platform. In a calm posture, the body is normally held upright and the center of mass is elevated above the base of support provided by the feet. Although it is generally assumed that the center of pressure (COP) indicates the location of the body's center of mass, discrepancies between the two occur, especially during rapid or high-frequency components of movement.
  Vestibular Dominant Score:indicates how much closing eyes and standing on a soft surface can affect the individual's ability to stand still and balanced.With eyes closed and on the mat, only the vestibular system is worked on and evaluated.The score will be calculated automatically by the device. Scoring ranges from 0 to 100. Higher scores are associated with better outcomes.
Gait Analysis(Step length) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Step length:During a gait cycle, the time from initial contact of one foot to initial contact of the opposite foot.Studies show a decrease in step length in people with MS compared to healthy controls. Pre- and post-intervention values will be compared
Gait Analysis(Stride length) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Stride length:the distance covered between the spot where one foot hits the ground and the next time that same foot hits the ground again.Studies show a decrease in stride length in people with MS compared to healthy controls. Pre- and post-intervention values will be compared
Gait Analysis(Step time) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Step time:the time from initial contact of one foot to initial contact of the opposite foot.The MS population displayed significantly longer step time in comparison to the healthy population.Pre- and post-intervention values will be compared
Gait Analysis(Step width) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Step width:Stride width is measured either between the medial-most borders of the two heels or between lines through the midline of the two heels. Normal stride width for adults is between 1-3 inches (3-8 cm). Stride width often increases with gait instability.The people with MS demonstrated a significantly increased step width when compared to healthy controls when walking at a self-selected pace in the literature.Pre- and post-intervention values will be compared
Gait Analysis(Cadence) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Cadence:is the number of steps taken per minute. People with the MS having a significantly reduced cadence in comparison to the healthy control population in the literature.Pre- and post-intervention values will be compared
Gait Analysis(Percentage distribution of walking phases) | 8th week
  The participants gait analysis will be performed using Diers pedogait. The participant will be asked to stand still on the treadmill at the beginning then walk of approximately 20 seconds at a speed chosen by the patient between 2-5 km/h. Diers pedoscan have been shown to be effective in detecting early-stage gait disorders in MS patients. Data to be evaluated after this measurement:
  Stance, Swing and Double support phase: The percentage ratios of the specified phases in a gait cycle will be calculated.In the literature, the MS population has significantly increased double support time when compared to the healthy control group. A significant increase in time spent in the swing phase was noted in the healthy population when compared to MS.Pre- and post-intervention values will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Sport Medicine Clinic, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsuda PN, Shumway-Cook A, Ciol MA, Bombardier CH, Kartin DA. Understanding falls in multiple sclerosis: association of mobility status, concerns about falling, and accumulated impairments. Phys Ther. 2012 Mar;92(3):407-15. doi: 10.2522/ptj.20100380. Epub 2011 Dec 1. PMID 22135709
- [Background] Martin CL, Phillips BA, Kilpatrick TJ, Butzkueven H, Tubridy N, McDonald E, Galea MP. Gait and balance impairment in early multiple sclerosis in the absence of clinical disability. Mult Scler. 2006 Oct;12(5):620-8. doi: 10.1177/1352458506070658. PMID 17086909
- [Background] Pollock AS, Durward BR, Rowe PJ, Paul JP. What is balance? Clin Rehabil. 2000 Aug;14(4):402-6. doi: 10.1191/0269215500cr342oa. PMID 10945424
- [Background] Prosperini L, Castelli L. Spotlight on postural control in patients with multiple sclerosis. Degener Neurol Neuromuscul Dis. 2018 Apr 3;8:25-34. doi: 10.2147/DNND.S135755. eCollection 2018. PMID 30050386
- [Background] Iqbal K. Mechanisms and models of postural stability and control. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:7837-40. doi: 10.1109/IEMBS.2011.6091931. PMID 22256156
- [Background] Creath R, Kiemel T, Horak F, Jeka JJ. The role of vestibular and somatosensory systems in intersegmental control of upright stance. J Vestib Res. 2008;18(1):39-49. PMID 18776597
- [Background] Melillo F, Di Sapio A, Martire S, Malentacchi M, Matta M, Bertolotto A. Computerized posturography is more sensitive than clinical Romberg Test in detecting postural control impairment in minimally impaired Multiple Sclerosis patients. Mult Scler Relat Disord. 2017 May;14:51-55. doi: 10.1016/j.msard.2017.03.008. Epub 2017 Mar 23. PMID 28619432
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Givon U, Zeilig G, Achiron A. Gait analysis in multiple sclerosis: characterization of temporal-spatial parameters using GAITRite functional ambulation system. Gait Posture. 2009 Jan;29(1):138-42. doi: 10.1016/j.gaitpost.2008.07.011. Epub 2008 Oct 31. PMID 18951800
- [Background] Thoumie P, Lamotte D, Cantalloube S, Faucher M, Amarenco G. Motor determinants of gait in 100 ambulatory patients with multiple sclerosis. Mult Scler. 2005 Aug;11(4):485-91. doi: 10.1191/1352458505ms1176oa. PMID 16042234
- [Background] Crenshaw SJ, Royer TD, Richards JG, Hudson DJ. Gait variability in people with multiple sclerosis. Mult Scler. 2006 Oct;12(5):613-9. doi: 10.1177/1352458505070609. PMID 17086908
- [Background] Gehlsen G, Beekman K, Assmann N, Winant D, Seidle M, Carter A. Gait characteristics in multiple sclerosis: progressive changes and effects of exercise on parameters. Arch Phys Med Rehabil. 1986 Aug;67(8):536-9. PMID 3741079
- [Background] Savci S, Inal-Ince D, Arikan H, Guclu-Gunduz A, Cetisli-Korkmaz N, Armutlu K, Karabudak R. Six-minute walk distance as a measure of functional exercise capacity in multiple sclerosis. Disabil Rehabil. 2005 Nov 30;27(22):1365-71. doi: 10.1080/09638280500164479. PMID 16372431
- [Background] Franceschini M, Rampello A, Bovolenta F, Aiello M, Tzani P, Chetta A. Cost of walking, exertional dyspnoea and fatigue in individuals with multiple sclerosis not requiring assistive devices. J Rehabil Med. 2010 Sep;42(8):719-23. doi: 10.2340/16501977-0600. PMID 20809053
- [Background] Gijbels D, Alders G, Van Hoof E, Charlier C, Roelants M, Broekmans T, Eijnde BO, Feys P. Predicting habitual walking performance in multiple sclerosis: relevance of capacity and self-report measures. Mult Scler. 2010 May;16(5):618-26. doi: 10.1177/1352458510361357. Epub 2010 Mar 5. PMID 20207785
- [Background] Hamilton F, Rochester L, Paul L, Rafferty D, O'Leary CP, Evans JJ. Walking and talking: an investigation of cognitive-motor dual tasking in multiple sclerosis. Mult Scler. 2009 Oct;15(10):1215-27. doi: 10.1177/1352458509106712. Epub 2009 Aug 10. PMID 19667011
- [Background] Langdon DW, Amato MP, Boringa J, Brochet B, Foley F, Fredrikson S, Hamalainen P, Hartung HP, Krupp L, Penner IK, Reder AT, Benedict RH. Recommendations for a Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). Mult Scler. 2012 Jun;18(6):891-8. doi: 10.1177/1352458511431076. Epub 2011 Dec 21. PMID 22190573
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Background] Strober LB, Rao SM, Lee JC, Fischer E, Rudick R. Cognitive impairment in multiple sclerosis: An 18 year follow-up study. Mult Scler Relat Disord. 2014 Jul;3(4):473-81. doi: 10.1016/j.msard.2014.03.004. Epub 2014 Apr 13. PMID 25877059
- [Background] Opara JA, Jaracz K, Brola W. Quality of life in multiple sclerosis. J Med Life. 2010 Oct-Dec;3(4):352-8. PMID 21254730
- [Background] das Nair R, Martin KJ, Lincoln NB. Memory rehabilitation for people with multiple sclerosis. Cochrane Database Syst Rev. 2016 Mar 23;3:CD008754. doi: 10.1002/14651858.CD008754.pub3. PMID 27004596
- [Background] Nasios G, Bakirtzis C, Messinis L. Cognitive Impairment and Brain Reorganization in MS: Underlying Mechanisms and the Role of Neurorehabilitation. Front Neurol. 2020 Mar 6;11:147. doi: 10.3389/fneur.2020.00147. eCollection 2020. PMID 32210905
- [Background] Motl RW, Sandroff BM, Benedict RH. Cognitive dysfunction and multiple sclerosis: developing a rationale for considering the efficacy of exercise training. Mult Scler. 2011 Sep;17(9):1034-40. doi: 10.1177/1352458511409612. Epub 2011 Jun 17. PMID 21685231
- [Background] Laver K, George S, Ratcliffe J, Crotty M. Virtual reality stroke rehabilitation--hype or hope? Aust Occup Ther J. 2011 Jun;58(3):215-9. doi: 10.1111/j.1440-1630.2010.00897.x. Epub 2011 Jan 9. No abstract available. PMID 21599688
- [Background] Lehrer N, Attygalle S, Wolf SL, Rikakis T. Exploring the bases for a mixed reality stroke rehabilitation system, part I: a unified approach for representing action, quantitative evaluation, and interactive feedback. J Neuroeng Rehabil. 2011 Aug 30;8:51. doi: 10.1186/1743-0003-8-51. PMID 21875441
- [Background] Beraud-Peigne N, Perrot A, Maillot P. Wireless Lighting System: A New Tool for Assessing Cognitive Functions in the Elderly. Behav Sci (Basel). 2023 Nov 17;13(11):943. doi: 10.3390/bs13110943. PMID 37998689
- [Background] Vasile AI, Stanescu MI. Strobe training as a visual training method that improves performance in climbing. Front Sports Act Living. 2024 May 20;6:1366448. doi: 10.3389/fspor.2024.1366448. eCollection 2024. PMID 38832310
- [Background] Ozakbas S, Yigit P, Cinar BP, Limoncu H, Kahraman T, Kosehasanogullari G. The Turkish validation of the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) battery. BMC Neurol. 2017 Dec 6;17(1):208. doi: 10.1186/s12883-017-0993-0. PMID 29207954
- [Background] Nortvedt MW, Riise T, Myhr KM, Nyland HI. Performance of the SF-36, SF-12, and RAND-36 summary scales in a multiple sclerosis population. Med Care. 2000 Oct;38(10):1022-8. doi: 10.1097/00005650-200010000-00006. PMID 11021675
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Trentzsch K, Schumann P, Sliwinski G, Bartscht P, Haase R, Schriefer D, Zink A, Heinke A, Jochim T, Malberg H, Ziemssen T. Using Machine Learning Algorithms for Identifying Gait Parameters Suitable to Evaluate Subtle Changes in Gait in People with Multiple Sclerosis. Brain Sci. 2021 Aug 7;11(8):1049. doi: 10.3390/brainsci11081049. PMID 34439668